CLINICAL TRIAL: NCT01931189
Title: A Clinical Pharmacokinetics Study of NI-071
Brief Title: Pharmacokinetics Study of NI-071
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nichi-Iko Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NI071A1
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NI-071 (Experimental)
  Interventions: Biological: NI-071
- Infliximab (Active Comparator)
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: NI-071 — 100mg/vial
  Arms: NI-071
Biological: Infliximab — 100mg/vial
  Other Names: Remicade
  Arms: Infliximab

SUMMARY:
The purpose of this study is to assess equivalence of pharmacokinetics between NI-071 and infliximab(the comparator) in Japanese healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, clinical laboratory tests, etc.)
2. Body Mass Index (BMI) of 18.5 to 25.0 kg/m2, and a total body weight of 50 to 80 kg

Exclusion Criteria:

1. Subjects with a following past History or concomitant diseases

   * Chronic or recurrent infectious disease
   * Demyelinating disease
   * Congestive heart failure
   * lymphoproliferative disorder or myelodysplastic syndrome
   * Malignancy
   * Interstitial lung disease
2. Subjects with active or latent tuberculosis or history of tuberculosis

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
PK : Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUCt) | 8 weeks

SECONDARY OUTCOMES:
PK : Area Under the Curve From Time Zero Extrapolated to Infinite Time (AUCinf) | 8 weeks
Safety : Incidence of Adverse Events | 8 weeks
Safety : Incidence of Anti-Drug Antibodies(ADA) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NichiIko Investigational Site, Tokyo, Japan